CLINICAL TRIAL: NCT05181800
Title: A Multi-center, Single-arm, Non-interventional Study to Describe the Safety of FIRMAGON® (Degarelix Acetate for Injection) in Chinese Patients With Prostate Cancer in Need of Androgen Deprivation Therapy
Brief Title: FIRMAGON® Intensive Drug Monitoring
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000351
Record Dates: First submitted 2021-12-20; First posted 2022-01-06 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FIRMAGON® Cohort
  Interventions: Other: Degarelix Cohort

INTERVENTIONS:
Other: Degarelix Cohort — Non-interventional
  Other Names: FIRMAGON®

SUMMARY:
To evaluate the safety profile of FIRMAGON® (to fulfill the regulatory authority's requirement of Intensive Drug Monitoring in Chinese participants with prostate cancer need androgen deprivation therapy [ADT] treated with FIRMAGON®).

Study Design

This study is a multi-center, single-arm, non-interventional, prospective study among Chinese participants with prostate cancer in need of ADT, receiving treatment with FIRMAGON®. This program provided the minimum 6 doses and maximum 12 doses of FIRMAGON® to enrolled participants during one-year follow-up. Participants who met the inclusion criteria would or were accepting at least 6 self-financed doses of treatment in a hospital. Participants should return to the hospital for medical assessment every three months. The prescription of 6 (3 doses × 2 times) self-financed doses will be given by doctors after assessment, and the direct-to-participant pharmacy will distribute FIRMAGON® to eligible participants (participants should bring the prescriptions and the last FIRMAGON® boxes to get other doses). All enrolled participants were followed up to collect safety information for one year from the 1st dose unless withdrawal of Informed Consent Form, discontinuation for 2 months, lost to follow-up, death, or termination due to other reasons, whichever came first.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer and in need of ADT
* Decision made to prescribe FIRMAGON® prior to enrollment
* Willingness and ability to provide written informed consent
* The participants are taking the marketed drug FIRMAGON®

Exclusion Criteria:

* Not signed informed consent
* Any participants who are unsuitable to participate in this study because of any other reasons will not be qualified to participate in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult participants with diagnosis of prostate cancer needing ADT.
Sampling Method: Non-Probability Sample
Enrollment: 1454 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- China Primary Healthcare Foundation, Beijing, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed at 145 investigational sites in China between August 2019 and December 2022.
Pre-assignment Details: In total, 1454 participants were screened and all the participants enrolled in the study
Groups:
- FIRMAGON Cohort: FIRMAGON Cohort: Non-interventional
Period: Overall Study
Arm/Group | FIRMAGON Cohort
Started | 1454
Completed | 1454
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FIRMAGON Cohort
Number analyzed (Participants) | 1454
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 300
  >=65 years | 1154
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1454
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1454
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 1454

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a medicinal product and which does not necessarily have to have a causal relationship with treatment.
Time Frame: From the signing of the informed consent up to the end-of-trial (12 months)
Measure: Count of Participants; unit: Participants
Arm/Group | FIRMAGON Cohort
Number analyzed (Participants) | 1454
Participants | 95

2. Primary Outcome: Percentage of Participants With Serious AEs
Description: An SAE was defined as any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or results in prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event or reaction.
Time Frame: From the signing of the informed consent up to the end-of-trial (12 months)
Measure: Count of Participants; unit: Participants
Arm/Group | FIRMAGON Cohort
Number analyzed (Participants) | 1454
Participants | 63

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent up to the end-of-trial (12 months)
Arm/Group | FIRMAGON Cohort
All-Cause Mortality (participants affected / at risk) | 55/1454
Serious Adverse Events (participants affected / at risk) | 63/1454
Other Adverse Events (participants affected / at risk) | 95/1454
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FIRMAGON Cohort (N=1454)
Pyrexia (General disorders) | 3 (3)
Injection site reactions (General disorders) | 2 (4)
Feeling cold (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Death (unknown cause) (General disorders) | 46 (46)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FIRMAGON Cohort (N=1454)
Pyrexia (General disorders) | 23 (30)
Injection site reactions (General disorders) | 17 (41)
Asthenia (General disorders) | 5 (5)
Chills (General disorders) | 3 (4)
Drug ineffective (General disorders) | 2 (2)
Feeling cold (General disorders) | 2 (2)
Feeling hot (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Marasmus (Metabolism and nutrition disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Urine abnormality (Renal and urinary disorders) | 1 (1)
Urinary tract inflammation (Renal and urinary disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Poor quality sleep (Psychiatric disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT05181800/Prot_SAP_000.pdf